CLINICAL TRIAL: NCT04394104
Title: COVID-19 Health and Wellness Self-Assessment Survey
Brief Title: COVID-19 Wellness Survey
Status: Terminated | Type: Observational
Why Stopped: Study has concluded.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Alexandra DelCollo, MS, MCHES, Senior Program Coordinator, Rutgers, The State University of New Jersey
Other Study IDs: Pro2020001009
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Survey Group: Group of individuals participating in the survey via self-selection. There is not intervention being administered. The group is simply answering questions on their health behaviors before COVID-19 and their health behaviors in the past 7-30 days, during the COVID-19 outbreak in the United States.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — No intervention is being administered.
  Other Names: There is no intervention

SUMMARY:
This study will collect data on physical activity, food consumption, stress, sleep, and alcohol consumption habits both before and after the national emergency for COVID-19 was put into place. This will help identify the health behavior changes taking place due to the COVID-19 pandemic in the United States. Data on past and current health behaviors will be self-reported by participants via a single online survey. The retrospective health behavior questions will be the same quantitative questions as the current health behavior questions so a direct comparison can be made. There will be a couple qualitative questions to assess what each participant feels are the greatest barriers or impacts to their current health behaviors. Participants will be recruited via convenient sampling.

Data collected in this study will show a decline in at least one healthy behavior after the United States national emergency for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Under the age of 18 and anyone who does not currently reside in the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Self-selected population
Sampling Method: Non-Probability Sample
Enrollment: 593 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Health Behavior Change Regression Questionnaire | 1-3 months
  A negative shift in health behaviors when comparing individual health behavior before COVID-19 and the last 7-30 days. This behavior change may be in one or multiple health behaviors measured. A negative shift is indicated by overall decrease in physical activity time or intensity, increase in sitting time, increase in alcohol consumption days or drinks on drinking occasions, a decrease in fruit/vegetable consumption, or indication of consuming more food.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers, The State University of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No